CLINICAL TRIAL: NCT01640613
Title: Anterior Approach Ultrasound-guided Intermediate Cervical Plexus Block for Carotid Endarterectomy
Brief Title: Anterior Ultrasound-guided Cervical Plexus Block for Carotid Endarterectomy
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Emmanuel Boselli, Md, PhD, Hôpital Edouard Herriot
Other Study IDs: 2012-A00147-36
Record Dates: First submitted 2012-07-06; First posted 2012-07-16 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Carotid Atherosclerosis; Regional Anesthesia Morbidity
Keywords: carotid endarterectomy; regional anaesthesia; ultrasound guided block
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe technique, efficiency, safety and satisfaction of ultrasound guided intermediate cervical plexus block for carotid endarterectomy.

The investigators present a simple approach for carotid regional anaesthesia by an anterior way that has not been published yet.

DETAILED DESCRIPTION:
* description of the anaesthetic procedure (duration, volume of anaesthetic local, efficiency)
* realization of the surgery (pain, injection of anaesthetic local...)
* post operative evaluation (pain, satisfaction...)

ELIGIBILITY:
Inclusion Criteria:

* adult
* carotid endarterectomy performed under regional anaesthesia

Exclusion Criteria:

* age < 18 years
* contralateral phrenic palsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing carotid endarterectomy under regional anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
conversion to general anaesthesia | surgery time

SECONDARY OUTCOMES:
amount of additional local anaesthetic | surgery time
  intraoperative supplementation by the surgeon
additional injection of remifentanil | surgery time
  In case of incontrolled pain : administration of remifentanil
complications | anaesthesia time
  hoarseness, Horner syndrome, cough, facial palsy
patient and surgeon satisfactions | after surgery
additional injection of remifentanil | surgery time
  In case of uncontrolled pain : administration of remifentanil

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Allaouchiche, MD PhD, Study Chair — Edouard Heriot Hospital, HCL; Emmanuel Boselli, MD PhD, Study Director — Edouard Heriot Hospital, HCL; Anne-Laure Calderon, MD, Principal Investigator — Edouard Heriot Hospital, HCL; Cyrille Truc, MD, Principal Investigator — Edouard Heriot Hospital, HCL; Julien Davidson, MD, Principal Investigator — Edouard Heriot Hospital, HCL; Najia Rahali, MD, Principal Investigator — Edouard Heriot Hospital, HCL; Farida Benatir, MD, Principal Investigator — Edouard Heriot Hospital, HCL
Locations (1):
- Departement of Anaesthesiology and Intensive Care, Edouard Heriot Hospital, HCL, Lyon, France